CLINICAL TRIAL: NCT04525547
Title: A Regulatory Required Non-interventional Study to Monitor the Safety and Effectiveness of Ofev(Nintedanib 150mg/100mg BID) in Korean Patients
Brief Title: Safety and Effectiveness of Nintedanib in Korean Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0417
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ofev treatment: Korean patients diagnosed with idiopathic pulmonary fibrosis, systemic sclerosis associated interstitial lung disease or chronic fibrosing interstitial lung diseases with a progressive phenotype receiving Ofev (nintedanib 150milligrams (mg)/100mg twice a day (BID))
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib
  Other Names: Ofev

SUMMARY:
The objectives of this study are to monitor the safety and effectiveness of Ofev in Korean patients in a routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been started on Ofev in accordance with the approved label in Korea
* Patients who have signed on the data release consent form

Exclusion Criteria:

* Patients for whom nintedanib is contraindicated according local label of Ofev

  * Patients with known hypersensitivity to Ofev, peanut or soya, or to any of the excipients
  * Women who are pregnant or nursing
  * Patients with moderate(Child pugh B) and severe(Child Pugh c) hepatic impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients diagnosed with idiopathic pulmonary fibrosis
  * (or) Patients diagnosed with systemic sclerosis associated interstitial lung disease
  * (or) patients diagnosed with chronic fibrosing ILD with a progressive phenotype
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- South Korea (22):
  - Dong-A University Hospital, Busan
  - Chungbuk national University Hospital, Chungcheongbuk-do
  - SoonChunHyang University Cheonan Hospital, Chungcheongnam-do
  - Keimyung University Dongsan Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Myongji Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gyeongsang National University Changwon Hospital, Gyeongsangnam-do
  - Jeju National University Hospital, Jeju-do
  - Wonkwang Univertisy Hospital, Jeollabuk-do
  - Jeonbuk National University Hospital, Jeollabuk-do
  - KyungHee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this non-interventional, multi-center study was to monitor the safety profile and effectiveness of Ofev in Korean patients diagnosed with idiopathic pulmonary fibrosis, systemic sclerosis associated interstitial lung disease or chronic fibrosing interstitial lung diseases with a progressive phenotype in routine clinical settings based on new collected data.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Ofev Treatment
Started | 70
Completed | 65
Not Completed | 5
Not completed — Not treated with Ofev | 2
Not completed — Off-label use | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all subjects who signed the data release consent form to participate in this study, took Ofev once at least, and were followed up by the physician once or more.
Arm/Group | Ofev Treatment
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.71 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Forced Vital Capacity (FVC) at baseline [Mean (Standard Deviation); unit: MilliLitres (mL)] — Population: The effectiveness set included safety set who were evaluated for the effectiveness including overall effectiveness evaluation.
  MilliLitres (mL)
    number analyzed (Participants) | 20
    (all) | 2510.00 (765.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events Who Took at Least One Dose of Ofev
Description: Number of patients with adverse events who took at least one dose of Ofev is presented.
Time Frame: Up to 24 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ofev Treatment
Number analyzed (Participants) | 65
Participants | 36

2. Primary Outcome: Change From Baseline in Forced Vital Capacity) (FVC) (mL) After 12 Weeks of Treatment
Description: Change from baseline in Forced Vital Capacity) (FVC) (mL) after 12 weeks of treatment is presented.
  Forced vital capacity (FVC) is part of a pulmonary function test that assesses the lung function. It is defined as the greatest volume of air that can be expelled when a person performs a rapid, forced exhalation.
Time Frame: At baseline and at week 12.
Population: The effectiveness set included safety set who were evaluated for the effectiveness including overall effectiveness evaluation. Only participants with non-missing results were included in the analysis.
Measure: Mean (Standard Deviation); unit: MilliLitres (mL)
Arm/Group | Ofev Treatment
Number analyzed (Participants) | 18
MilliLitres (mL) | -15.00 (270.73)
Statistical Analysis 1: Comparison: Ofev Treatment; Test type: Other; p = 0.8170, t-test, 2 sided

3. Primary Outcome: Change From Baseline in Forced Vital Capacity) (FVC) (mL) After 24 Weeks of Treatment
Description: Change from baseline in Forced Vital Capacity) (FVC) (mL) after 24 weeks of treatment is presented.
  Forced vital capacity (FVC) is part of a pulmonary function test that assesses the lung function. It is defined as the greatest volume of air that can be expelled when a person performs a rapid, forced exhalation.
Time Frame: At baseline and at week 24.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: MilliLitres (mL)
Arm/Group | Ofev Treatment
Number analyzed (Participants) | 10
MilliLitres (mL) | -44.00 (299.49)
Statistical Analysis 1: Comparison: Ofev Treatment; Test type: Other; p = 0.6533, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 24 weeks.
Description: The safety set included all subjects who signed the data release consent form to participate in this study, took Ofev once at least, and were followed up by the physician once or more.
Arm/Group | Ofev Treatment
All-Cause Mortality (participants affected / at risk) | 3/65
Serious Adverse Events (participants affected / at risk) | 16/65
Other Adverse Events (participants affected / at risk) | 17/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofev Treatment (N=65)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
COVID-19 (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Asthenia (General disorders) | 1
Generalised oedema (General disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Weight decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofev Treatment (N=65)
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04525547/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT04525547/SAP_001.pdf